CLINICAL TRIAL: NCT04864587
Title: Artificial Intelligence in Image Recognition of Pouchoscopies in Patients With Restorative Proctocolectomy
Acronym: PouchVision
Status: Completed | Type: Observational
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: PouchVision1.0
Record Dates: First submitted 2021-04-21; First posted 2021-04-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pouches, Ileoanal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Restorative colectomy with ileoanal pouch: Patients with restorative colectomy with ileoanal pouch who receive pouchoscopy for detection of pouchitis or neoplasm
  Interventions: Diagnostic Test: Artificial intelligence used for image recognition in pouchoscopy

INTERVENTIONS:
Diagnostic Test: Artificial intelligence used for image recognition in pouchoscopy — The aim of this study is to develop an image recognition algorithm that reliably detects the different graduations of pouch inflammation and neoplasms in the pouch

SUMMARY:
The application of artificial intelligence in pouchoscopy of patients with restorative proctocolectomy might improve the diagnosis of pouchitis and neoplasms. The aim of this pilot study is to develop a convolutional neural network algorithm for pouchoscopy

DETAILED DESCRIPTION:
Restorative proctocolectomy is the standard procedure for treatment of refractory severe colitis in inflammatory bowel disease as well as the standard procedure for carcinoma preventive treatment of patients with inflammatory bowel disease with colonic neoplasia and patients with familial adenomatous polyposis coli (FAP). Pouchoscopy can be used to monitor the success of therapy and to detect complications such as pouchitis or neoplasia. Artificial Intelligence assisted image recognition programs can support the examiner in finding a diagnosis and train physicians in training, objectify endoscopic findings in the context of studies and might make biopsies unnecessary, thus saving costs. The application of Artificial Intelligence in pouchoscopy has not been demonstrated to date. The aim of this study is to develop, an image recognition algorithm that reliably detects the different graduations of pouch inflammation. This requires training and fine-tuning of the image recognition program PiTorch using the largest possible amount of image data, which will be recruited from the image databases of the UMM and the Theresienkrankenhaus Mannheim. A test run for statistical evaluation will be performed on an independent cohort.

ELIGIBILITY:
Inclusion Criteria:

• All patients aged ≥ 18 years with inflammatory bowel disease and status after restorative proctocolectomy with ileoanal pouch who had received a pouchoscopy

Exclusion Criteria:

• Very poor endoscopic image quality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with inflammatory bowel disease and status after restorative proctocolectomy with ileoanal pouch might develop pouchitis or neoplasia in the pouch.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
AI versus endoscopist | Immediately after application of AI algorithm or after assessment of the endoscopic image by the endoscopist
  Detection of pouchitis by AI versus assessment by endoscopist in pouchoscopy
AI versus pathologist | Immediately after application of AI algorithm or after assessment of the microscopic image of the pouch biopsy by the pathologist
  Detection of pouchitis by AI versus pathologist in pouchoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, PhD, Principal Investigator — Theresienkrankenhaus Mannheim, University of Heidelberg
Locations (1):
- Theresienkrankenhaus und St. Hedwigkliniken GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Sommen F, de Groof J, Struyvenberg M, van der Putten J, Boers T, Fockens K, Schoon EJ, Curvers W, de With P, Mori Y, Byrne M, Bergman JJGHM. Machine learning in GI endoscopy: practical guidance in how to interpret a novel field. Gut. 2020 Nov;69(11):2035-2045. doi: 10.1136/gutjnl-2019-320466. Epub 2020 May 11. PMID 32393540